CLINICAL TRIAL: NCT01964560
Title: A Multicenter, Open-label, Long-term Extension Study to Investigate the Efficacy and Safety of Lacosamide as Adjunctive Therapy in Pediatric Subjects With Epilepsy With Partial-Onset Seizures
Brief Title: A Clinical Study to Investigate the Efficacy and Safety of Lacosamide as an Add on Therapy in Children With Epilepsy With Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Collaborators: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EP0034; 2012-005012-26 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy
Keywords: Lacosamide; Vimpat; UCB; Epilepsy; Partial-Onset Seizures; Pediatric
MeSH Terms: conditions — Epilepsy | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): In the first week after enrollment into EP0034 subjects will be dosed according to their weight:
  * Lacosamide (LCM) 10 mg/kg/day (oral solution) for subjects weighing <30 kg
  * LCM 6 mg/kg/day (oral solution) for subjects weighing ≥30 kg to <50 kg
  * LCM 300 mg/day (tablets) for subjects weighing ≥50 kg
  After 1 week the investigator may adjust the LCM dose during the Treatment Period based on clinical judgment within a range of 2 mg/kg/day to 12 mg/kg/day for the oral solution and 100 mg/day to 600 mg/day for the tablets.
  Interventions: Drug: Lacosamide

INTERVENTIONS:
Drug: Lacosamide — Pharmaceutical form: oral solution
  Concentration: 1 mg/kg - 6 mg/kg BID (2 mg/kg/day - 12 mg/ kg/day)
  Route of administration: oral use
  Other Names: VIMPAT
Drug: Lacosamide — Pharmaceutical form: tablet
  Concentration: 50 mg - 300 mg BID (100 mg/day - 600 mg/day)
  Route of administration: oral use
  Other Names: VIMPAT

SUMMARY:
The purpose of this study is to evaluate the long-term safety, tolerability and efficacy of lacosamide (LCM) in pediatric subjects.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written Informed Consent form (ICF) is signed and dated by the subject or legal representative. The ICF or a specific Assent form, where required, will be signed and dated by minors
* Subject has completed the Transition Period of SP0967 [NCT02477839] or SP0969 [NCT01921205] for the treatment of uncontrolled partial-onset seizures in pediatric epilepsy
* Subject is expected to benefit from participation, in the opinion of the investigator
* Subject/legal representative is considered reliable and capable of adhering to the protocol (eg, able to understand and complete diaries), visit schedule, and medication intake according to the judgment of the investigator
* Subject is male or female aged 1 month to ≤17 years
* Subject has a diagnosis of epilepsy with partial-onset seizures

Exclusion Criteria:

* Subject is receiving any investigational drugs or using any experimental devices in addition to lacosamide (LCM)
* Subject meets a mandatory withdrawal criterion (ie, MUST withdraw criterion) for SP0967 or SP0969, or is experiencing an ongoing serious adverse event (SAE)
* For subjects ≥6 years of age, subject has a lifetime history of suicide attempt (including an actual attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ('Yes') to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Visit 1
* Female subject who is pregnant or nursing, and/or a female subject of childbearing potential who is not surgically sterile or does not practice 1 highly effective method of contraception

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 540 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (141):
- United States (11):
  - Ep0034 638, Birmingham, Alabama
  - Ep0034 105, Orlando, Florida
  - Ep0034 117, Tampa, Florida
  - Ep0034 124, Lexington, Kentucky
  - Ep0034 115, Henderson, Nevada
  - Ep0034 120, Lebanon, New Hampshire
  - Ep0034 102, Charlotte, North Carolina
  - Ep0034 640, Springfield, Oregon
  - Ep0034 129, Dallas, Texas
  - Ep0034 630, San Antonio, Texas
  - Ep0034 114, Seattle, Washington
- Argentina (2):
  - Ep0034 143, Ciudad Autonoma de Buenos AIRE
  - Ep0034 142, Córdoba
- Australia (3):
  - Ep0034 200, Melbourne
  - Ep0034 203, Parkville
  - Ep0034 205, South Brisbane
- Ep0034 304, Brussels, Belgium
- Brazil (3):
  - Ep0034 158, Passo Fundo
  - Ep0034 150, São Paulo
  - Ep0034 154, São Paulo
- Ep0034 310, Plovdiv, Bulgaria
- China (6):
  - Ep0034 530, Beijing
  - Ep0034 535, Changchun
  - Ep0034 532, Chongqing
  - Ep0034 536, Nanchang
  - Ep0034 531, Shanghai
  - Ep0034 537, Shenzhen
- Ep0034 171, Medellín, Colombia
- Croatia (3):
  - Ep0034 613, Osijek
  - Ep0034 610, Rijeka
  - Ep0034 612, Zagreb
- Czechia (4):
  - Ep0034 321, Hradec Králové
  - Ep0034 320, Ostrava-poruba
  - Ep0034 323, Prague
  - Ep0034 322, Praha 4 - KRC
- Estonia (2):
  - Ep0034 331, Tallinn
  - Ep0034 330, Tartu
- France (2):
  - Ep0034 346, Rennes
  - Ep0034 344, Strasbourg
- Georgia (4):
  - Ep0034 620, Tbilisi
  - Ep0034 621, Tbilisi
  - Ep0034 622, Tbilisi
  - Ep0034 623, Tbilisi
- Ep0034 542, Athens, Greece
- Hungary (8):
  - Ep0034 361, Budapest
  - Ep0034 362, Budapest
  - Ep0034 363, Budapest
  - Ep0034 364, Budapest
  - Ep0034 368, Budapest
  - Ep0034 360, Debrecen
  - Ep0034 367, Miskolc
  - Ep0034 366, Pécs
- Ep0034 374, Petah Tikva, Israel
- Italy (9):
  - Ep0034 397, Genova
  - Ep0034 380, Mantova
  - Ep0034 398, Messina
  - Ep0034 381, Milan
  - Ep0034 393, Padua
  - Ep0034 383, Roma
  - Ep0034 392, Roma
  - Ep0034 395, Roma
  - Ep0034 386, Verona
- Latvia (2):
  - Ep0034 400, Riga
  - Ep0034 402, Valmiera
- Ep0034 411, Kaunas, Lithuania
- Mexico (6):
  - Ep0034 694, Aguascalientes
  - Ep0034 569, Culiacán
  - Ep0034 693, Culiacán
  - Ep0034 563, Guadalajara
  - Ep0034 564, México
  - Ep0034 568, Monterrey
- Ep0034 650, Chisinau, Moldova
- Ep0034 660, Podgorica, Montenegro
- Philippines (2):
  - Ep0034 724, Cebu
  - Ep0034 721, Manila
- Poland (9):
  - Ep0034 433, Gdansk
  - Ep0034 420, Kielce
  - Ep0034 422, Krakow
  - Ep0034 431, Krakow
  - Ep0034 423, Poznan
  - Ep0034 425, Poznan
  - Ep0034 429, Tyniec Mały
  - Ep0034 430, Warsaw
  - Ep0034 428, Wroclaw
- Ep0034 750, Lisbon, Portugal
- Romania (9):
  - Ep0034 574, Bucharest
  - Ep0034 581, Bucharest
  - Ep0034 572, Cluj-Napoca
  - Ep0034 582, Iași
  - Ep0034 573, Sibiu
  - Ep0034 576, Sibiu
  - Ep0034 580, Suceava
  - Ep0034 570, Timișoara
  - Ep0034 577, Timișoara
- Russia (16):
  - Ep0034 443, Kazan'
  - Ep0034 444, Kazan'
  - Ep0034 454, Kemerovo
  - Ep0034 442, Moscow
  - Ep0034 449, Moscow
  - Ep0034 456, Nizhny Novgorod
  - Ep0034 452, Novosibirsk
  - Ep0034 453, Omsk
  - Ep0034 455, Perm
  - Ep0034 441, Saint Petersburg
  - Ep0034 446, Saint Petersburg
  - Ep0034 440, Smolensk
  - Ep0034 730, Smolensk
  - Ep0034 458, Tomsk
  - Ep0034 447, Voronezh
  - Ep0034 450, Yekaterinburg
- Serbia (5):
  - Ep0034 461, Belgrade
  - Ep0034 464, Belgrade
  - Ep0034 460, Kragujevac
  - Ep0034 462, Novi Sad
  - Ep0034 463, Novi Sad
- Slovakia (2):
  - Ep0034 470, Bardejov
  - Ep0034 472, Nové Zámky
- Ep0034 670, Ljubljana, Slovenia
- South Korea (5):
  - Ep0034 211, Daegu
  - Ep0034 210, Seoul
  - Ep0034 212, Seoul
  - Ep0034 213, Seoul
  - Ep0034 215, Seoul
- Taiwan (3):
  - Ep0034 220, Changhua
  - Ep0034 222, Taichung
  - Ep0034 224, Taipei
- Thailand (6):
  - Ep0034 236, Bangkoknoi
  - Ep0034 235, Pathum Wan
  - Ep0034 230, Ratchathewi
  - Ep0034 232, Ratchathewi
  - Ep0034 231, Tha Muang
  - Ep0034 233, Tha Muang
- Ukraine (7):
  - Ep0034 602, Dnipro
  - Ep0034 609, Dnipro
  - Ep0034 681, Ivano-Frankivsk
  - Ep0034 600, Kiev
  - Ep0034 606, Kiev
  - Ep0034 682, Uzhhorod
  - Ep0034 603, Vinnytsia
- United Kingdom (2):
  - Ep0034 515, Cambridge
  - Ep0034 511, Leeds

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- See also: Product Information — https://www.ucb.com/_up/ucb_com_products/documents/Vimpat_Labeling_Oct_2021.pdf
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in August 2014 and concluded in April 2022.
Pre-assignment Details: The Participant Flow refers to the Safety Set (SS). The SS included all enrolled study participants who took at least 1 dose of lacosamide (LCM) in this long-term extension study.
Groups:
- Lacosamide (All Subjects): Participants who participated in primary study [SP0967 (NCT02477839) or SP0969 (NCT01921205)] consented and met requirements to participate in current study received LCM 10 milligram/kilogram/day (mg/kg/day) as an oral solution for study participants weighing <30 kg, LCM 6 mg/kg/day as an oral solution for study participants weighing >=30 kg to <50 kg, and LCM 300 mg/day as tablets for study participants weighing >=50 kg. LCM was administered twice daily (bid) up to Week 96. After 1 week the investigator might adjust the LCM dose during the Treatment based on clinical judgment within a range of 2 mg/kg/day to 12 mg/kg/day for the oral solution and 100 mg/day to 600 mg/day for the tablets.
Period: Overall Study
Arm/Group | Lacosamide (All Subjects)
Started | 540
Completed | 395
Not Completed | 145
Not completed — Adverse Event | 23
Not completed — Lack of Efficacy | 46
Not completed — Protocol deviation | 2
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 64
Not completed — Surgery-hemispherotomy | 1
Not completed — Surgery | 1
Not completed — Seizures appeared resolved with epilepsy surgery | 1
Not completed — Patient and Investigator choice | 1
Not completed — Patient was prescribed CBD | 1
Not completed — Participant moved to another country | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all enrolled study participants who took at least 1 dose of LCM in this long-term extension study.
Arm/Group | Lacosamide (All Subjects)
Number analyzed (Participants) | 540
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.486 (5.415)
Age, Customized [Count of Participants; unit: Participants]
  >=28 days - <24 months | 103
  >=24 months - <12 years | 287
  >=12 - <18 years | 150
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236
  Male | 304
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan native | 18
  Asian | 83
  Black | 4
  White | 414
  Other/mixed | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 68
  Not Hispanic or Latino | 472

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. Treatment-emergent is defined as starting on or after the date of first dose of LCM in EP0034, and within 30 days of last dose.
Time Frame: From Week 0 to the End of Safety Follow-Up (up to Week 104)
Population: The Safety Set (SS) included all enrolled study participants who took at least 1 dose of LCM in this long-term extension study.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide (All Subjects)
Number analyzed (Participants) | 540
percentage of participants | 77.2

2. Primary Outcome: Percentage of Participants With Serious TEAEs
Description: A serious adverse event (SAE) must meet 1 or more of the following criteria: • Death, • Life-threatening (Life-threatening does not include a reaction that might have caused death had it occurred in a more severe form.), • Significant or persistent disability/incapacity, • Congenital anomaly/birth defect (including that occurring in a fetus), • Important medical event that, based upon appropriate medical judgment, may jeopardize the patient or participant and may require medical or surgical intervention to prevent 1 of the other outcomes listed in the definition of serious., • Initial inpatient hospitalization or prolongation of hospitalization. Treatment-emergent is defined as starting on or after the date of first dose of LCM in EP0034, and within 30 days of last dose.
Time Frame: From Week 0 to the End of Safety Follow-Up (up to Week 104)
Population: The SS included all enrolled study participants who took at least 1 dose of LCM in this long-term extension study.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide (All Subjects)
Number analyzed (Participants) | 540
percentage of participants | 20.6

3. Primary Outcome: Percentage of Participants With TEAEs Leading to Study Discontinuation
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. AEs leading to study discontinuation. Treatment-emergent is defined as starting on or after the date of first dose of LCM in EP0034, and within 30 days of last dose.
Time Frame: From Week 0 to the End of Safety Follow-Up (up to Week 104)
Population: The SS included all enrolled study participants who took at least 1 dose of LCM in this long-term extension study. Here, only those participants who discontinued the study due to TEAEs starting on or after the date of first dose of LCM in EP0034, and within 30 days of last dose of LCM are reported.
Measure: Number; unit: percentage of participants
Arm/Group | Lacosamide (All Subjects)
Number analyzed (Participants) | 540
percentage of participants | 4.1

4. Secondary Outcome: Percentage of Seizure-free Days During the Study
Description: The number of seizure-free days was the total number of days within an interval for which daily diary data were available and no seizures were reported. The percentage of seizure-free days was computed as 100 times the number of seizure-free days in the interval divided by the number of days in the interval for which daily diary data were available. Percentage of seizure-free days was measured using data obtained from participant diaries from EP0034 and is presented for the overall Treatment only.
Time Frame: From Week 0 to End of Treatment (up to Week 96)
Population: The Full Analysis Set (FAS) was used for the analysis of seizure data and included all study participants in the SS who had at least 1 completed post-Baseline seizure diary. Study participants whose efficacy data could not be source verified were excluded from the FAS. Here, Number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Mean (Standard Deviation); unit: percentage of seizure free days
Arm/Group | Lacosamide (All Subjects)
Number analyzed (Participants) | 537
percentage of seizure free days | 66.96 (36.18)

ADVERSE EVENTS:
Time Frame: From Week 0 to the End of Safety Follow-Up (up to Week 104)
Description: TEAEs were events which started on or after date of first EP0034 dose of LCM, or whose intensity worsened on or after date of first EP0034 dose of LCM. AEs occurring within 30 days after last dose of LCM were considered treatment-emergent. SS included all enrolled study participants who took at least 1 dose of LCM in the long-term extension study.
Arm/Group | Lacosamide (All Subjects)
All-Cause Mortality (participants affected / at risk) | 7/540
Serious Adverse Events (participants affected / at risk) | 111/540
Other Adverse Events (participants affected / at risk) | 289/540
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (All Subjects) (N=540)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cerebral palsy (Congenital, familial and genetic disorders) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 1 (2)
Blepharitis (Eye disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Parophthalmia (Eye disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (12)
Nausea (Gastrointestinal disorders) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Device malfunction (General disorders) | 2 (3)
Cyst (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Device breakage (General disorders) | 1 (1)
Device occlusion (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 11 (14)
Bronchitis (Infections and infestations) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 4 (5)
Bronchopneumonia (Infections and infestations) | 3 (4)
Dengue fever (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 2 (2)
Influenza (Infections and infestations) | 2 (2)
Rhinovirus infection (Infections and infestations) | 2 (2)
Abscess neck (Infections and infestations) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1)
Amoebic dysentery (Infections and infestations) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Enterovirus infection (Infections and infestations) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
Viral infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Post procedural fistula (Injury, poisoning and procedural complications) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Acetonaemia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Enteral feeding intolerance (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (2)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1)
Convulsion (Nervous system disorders) | 24 (30)
Status epilepticus (Nervous system disorders) | 9 (11)
Epilepsy (Nervous system disorders) | 7 (10)
Partial seizures (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 3 (3)
Partial seizures with secondary generalisation (Nervous system disorders) | 3 (5)
Febrile convulsion (Nervous system disorders) | 2 (2)
Hemiparesis (Nervous system disorders) | 2 (2)
Somnolence (Nervous system disorders) | 2 (3)
Altered state of consciousness (Nervous system disorders) | 1 (2)
Cognitive disorder (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1)
Intracranial haematoma (Nervous system disorders) | 1 (1)
Motor dysfunction (Nervous system disorders) | 1 (1)
Myoclonic epilepsy (Nervous system disorders) | 1 (1)
Subdural hygroma (Nervous system disorders) | 1 (1)
Tonic convulsion (Nervous system disorders) | 1 (1)
Disorientation (Psychiatric disorders) | 1 (1)
Emotional disorder of childhood (Psychiatric disorders) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (2)
Pyuria (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 1 (1)
Brain operation (Surgical and medical procedures) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (All Subjects) (N=540)
Vomiting (Gastrointestinal disorders) | 56 (113)
Diarrhoea (Gastrointestinal disorders) | 42 (54)
Pyrexia (General disorders) | 86 (149)
Upper respiratory tract infection (Infections and infestations) | 83 (167)
Nasopharyngitis (Infections and infestations) | 57 (92)
Pharyngitis (Infections and infestations) | 39 (68)
Bronchitis (Infections and infestations) | 33 (46)
Influenza (Infections and infestations) | 28 (35)
Somnolence (Nervous system disorders) | 30 (42)
Headache (Nervous system disorders) | 29 (89)
Convulsion (Nervous system disorders) | 27 (33)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-11-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT01964560/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-03): https://cdn.clinicaltrials.gov/large-docs/60/NCT01964560/SAP_001.pdf